CLINICAL TRIAL: NCT01820338
Title: Extension Family Lifestyle Intervention Project (E-FLIP for Kids)
Acronym: E-FLIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 204-2009
Record Dates: First submitted 2013-03-19; First posted 2013-03-28 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Obesity
Keywords: Children, Obesity, Intervention
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Behavioral Family Intervention (Experimental): Child and Parent attend intervention including nutrition and physical activity education, plus behavioral strategies to facilitate behavior and weight status change
  Interventions: Behavioral: Behavioral Child Tx Contacts; Behavioral: Behavioral Parent-Tx Contacts; Other: Dietary and Physical Activity Information
- Behavioral Parent-Only Intervention (Experimental): Only parents attend intervention including nutrition and physical activity education, plus behavioral strategies to facilitate behavior and weight status change
  Interventions: Behavioral: Behavioral Parent-Tx Contacts; Other: Dietary and Physical Activity Information
- Education Control (Active Comparator): Child and parent attend intervention that includes only nutrition and physical activity education; no instruction or assistance in the use of behavioral strategies are included in this condition
  Interventions: Other: Dietary and Physical Activity Information

INTERVENTIONS:
Behavioral: Behavioral Child Tx Contacts — Each parent and child dyad will participate in group meetings. Children and parents will meet in simultaneous, but separate, groups at each meeting. The intervention will include 12 sessions over 16 weeks. Families will also participate in a maintenance intervention for the next eight months. The primary treatment objectives will be to decrease caloric intake in a nutritionally sound manner and to increase moderate intensity exercise. Changes in dietary habits will be addressed via a modified version of the Stoplight System. Children and adults will be encouraged to eat a well-balanced diet based on the food guide pyramid. Parents and children will also be given pedometers and they will be asked to keep track of the number of steps they take each day. Each week parents and children will set goals to gradually increase physical activity. Parent and their children will be asked to record what they eat and drink, as well as their physical activity on daily food logs.
  Arms: Behavioral Family Intervention
Behavioral: Behavioral Parent-Tx Contacts — Only the participating parent(s) will attend group meetings. The intervention will include weekly sessions for the first 8 weeks and biweekly sessions for the next 8 weeks. They will also participate in a maintenance intervention for eight months. Each session will last 90 minutes. The sessions for parents in the parent-only program will be structured the same as the parents sessions for the family-based intervention and will also cover the same topics. As with the family-based intervention, the parent and their children assigned to the parent-only intervention will be asked to record what they eat and drink, as well as their physical activity, on a daily basis. Each week group interventionists will model the goal setting process with parents and suggest a general range of age-appropriate dietary and physical activity targets that might be appropriate for each child and parent.
  Arms: Behavioral Family Intervention; Behavioral Parent-Only Intervention
Other: Dietary and Physical Activity Information — Both the child and parent will attend the treatment sessions in this program. The condition will include a series of meetings addressing key aspects of nutrition, physical activity, and health promotion such as national guidelines regarding proper nutrition, guidelines for physical activity, strategies to cope with stress, healthy sources and guidelines for intake of fiber, calcium, protein, grains & carbohydrates. Topics will also include use of vitamin & mineral supplements, dental and sleep hygiene, self-esteem, family communication, and assertiveness training in dealing with peer victimization. The families in the Health Education group will not receive training in behavioral self-regulation strategies, such as goal setting and self-monitoring. Children will participate in a group physical activity during each session such as frisbee, jump rope, stoplight tag. They will also sample healthy snacks such as pretzels or fruits and vegetables.

SUMMARY:
The Extension Family Lifestyle Intervention Project (E-FLIP for Kids) trial will evaluate the impact of a community based intervention delivered to families in rural settings utilizing the existing Cooperative Extension Service network on child dietary intake and weight. Specifically, the E-FLIP for Kids study will determine if behavioral treatments for child obesity lead to greater improvement in child weight compared to educational only treatment.Participants will include 240 parent-child dyads from ten rural counties in north central Florida. Study outcomes will be measure prior to treatment, at the end of treatment (month 12) and at one year follow-up (month 24). All treatment meetings will be held at Cooperative Extension Service offices within each participating county.

DETAILED DESCRIPTION:
The study sample will include 240 overweight and obese children, ages 8 to 12 years, and their parent(s) from rural counties in North Central Florida. Participants will be randomized to one of three conditions: family-based (FB) healthy lifestyle intervention, parent-only (PO) healthy lifestyle intervention, and health education control (HEC) condition. Each of the treatment conditions will involve 23 group meetings delivered on the same schedule.

Recruitment will include direct solicitation methods combined with culturally-tailored efforts targeting the recruitment of minority participants. Direct solicitation methods will entail direct mailings to households and to health-care providers, a press release, and presentations/brochure distribution by Extension agents and research team members at churches, social organizations, community events, and through local businesses. Brochures will also be distributed through local schools. Recruitment information will contain a toll-free phone number to our research office. Potential participants will be encouraged to call our office to learn more about the study and complete an initial phone screen. The phone calls will be received by trained staff that will describe the study and perform a brief phone screen in order to determine initial eligibility. Those families who meet initial eligibility and express interest will be scheduled for an in-person screening visit to determine their final eligibility for the program.

Participants (child and parent) will complete assessment measures at an initial screening visit, pre-start baseline assessment, post-treatment assessment (12 months after the baseline assessment), and a follow-up assessment (24 months after the baseline assessment).

At the initial in-person screening visit interested participants (child and parent/legal guardian) will complete informed consent procedures and then measures of height and weight, medical history questionnaires, and a general family information form. Parents will complete questionnaires regarding family functioning, parent psychological functioning, parent mobility, child behavior, reasons for seeking treatment, and family cost of program participation. Children will complete questionnaires regarding reasons for joining the program and social interactions. In addition, the child will be assessed for resting heart rate and blood pressure.

The pre-start/baseline assessment visit will occur approximately one to two weeks prior to the beginning of the intervention. At this assessment children and parents will be measured for height and weight, and the child's waist circumference will also be assessed. Families will complete a packet of self-report study questionnaires. Children will be assessed for blood pressure and heart rate. Children's body fat percentage will be assessed by an electrical impedence scale. Child will be asked to wear an armband accelerometer for seven days following the assessment. Children will also be asked to complete one finger prick (with collection of approximately 2-3 drops of blood) to assess blood lipids and HbA1C using a point-of-care device. A 20 meter shuttle physical fitness assessment will also be completed by children to assess their level of physical fitness. The finger prick, blood pressure, physical fitness, and heart rate assessment protocol will be completed by study medical personnel trained in these procedures. Children, with help from their parents, will complete measures of the child's dietary intake and physical activity habits, eating behaviors, qualify of life, body image, and pubertal development. Parents will complete measures about their own dietary intake and physical activity habits, the family feeding environment, perceive family support and social problem solving abilities. At the end of this baseline assessment visit, participants will be notified as to which of the three treatment conditions they were randomized.

The same assessment protocol administered at the baseline visit will be administered at the post-treatment assessment, and follow-up assessment. Measures of post-treatment satisfaction will also be administered to the child and parent at these two follow-up assessments.

Family-Based Group Intervention Condition: Each parent and child dyad will participate in 23 group meetings. Children and parents will meet in simultaneous, but separate, parent and child groups at each meeting. The intervention will include weekly sessions for the first 8 weeks and biweekly sessions for the next 8 weeks. Families will also participate in a maintenance intervention for the next eight months (months 5 to 12) that includes one session per month, with the exception of month 8, which will include 4 weekly sessions. For all child and parent participants, the primary treatment objectives will be to decrease caloric intake in a nutritionally sound manner and to increase moderate intensity exercise. Changes in dietary habits will be addressed via a modified version of the Stoplight System. The stoplight system is designed to teach children and parents to classify foods according to the colors of the stoplight. Green foods are "go foods", are foods high in nutrients and low in calories (i.e., fruits and vegetables). Yellow foods are "caution" foods. Yellow foods have lots of nutrition, but also significant calories and should be eaten in moderation. Red foods are "stop" foods. These foods are high in calories relative to nutrients. Red foods should be limited, but are not considered forbidden. Weekly goals will target gradual reductions in caloric intake through limiting consumption of high-fat/high-sugar foods "Red foods" and increasing consumption of fruits and vegetables. Children and adults will be encouraged to eat a well-balanced diet based on the food guide pyramid. Parents and children will also be given pedometers (step counters) and they will be asked to keep track of the number of steps they take each day. Each week parents and children will set goals to gradually increase the number of steps they take each day. Parent and their children will be asked to record what they eat and drink, as well as their physical activity (number of steps taken) on daily food logs.

Parent Group Session. Each session will last 90 minutes and will include three segments. In the first segment will review parent and child progress in implementing the strategies recommended and goals set for changing their eating or exercise in the previous session. Parents will discuss with group leaders the successes, challenges, and barriers encountered as they attempted to make lifestyle changes over the past week, as well as discuss possible strategies for overcoming various challenges. The second segment will focus on the specific "topic of the day" or "session lesson". The third segment will involve bringing the children and parents back together at the end of each session to set specific goals for the next week.

Child Group Session. Each session will last 90 minutes. During the first part of the session we will review the children's progress in achieving their dietary and physical activity goals over the previous week. After a private weigh-in, child participants will describe the progress they achieved in reaching their dietary and physical activity goals. Good progress will be highlighted by strong positive feedback. The second segment will include an exercise or game component to demonstrate strategies/activities to help children keep physically active including activities such as Frisbee, flashlight tag, watermelon relay, jump rope, kickball and dancing. Third, the children and group leaders will prepare and sample a variety of healthy snacks including fruits and vegetables with various healthy low fat dips, bagels with low fat cream cheese, low fat cheese quesadillas, fruit smoothies, and yogurt fruit parfaits. During the food sampling portion of each session, fun and educational activities will be used to teach children about nutrition (e.g., recognizing calorie and fat content of foods via "signals" of the Stoplight program), strategies to increase physical activity, behavioral management skills (self-monitoring and goal setting), and strategies to cope with psychosocial concerns (i.e., building self-esteem) and how to also support their parents.

Parent-only Group Intervention Condition: Only the participating parent(s) will attend 23 group meetings over the course of one year. The parent-only interventions will meet on the same schedule as the family-based intervention. The intervention will include weekly sessions for the first 8 weeks and biweekly sessions for the next 8 weeks. Families will also participate in a maintenance intervention for eight months (months 5 to 12) that includes one session per month, with the exception of month 8, which will include 4 weekly sessions.

Each session will last 90 minutes and will include three segments, similar to the parent group previously described in the FB intervention. The sessions for parents in the parent-only program will be structured the same as the parents sessions for the family-based intervention (described above) and will also cover the same topics. As with the family-based intervention, the parent and their children assigned to the parent-only intervention will be asked to record what they eat and drink, as well as their physical activity, on a daily basis. As children will not be attending group sessions in this condition, an emphasis will be placed on helping parents effectively communicate the topics of each session to the target child at home, as well as teaching parents how to work with their children to set goals together and monitor their food intake and physical activity. Each week group interventionists will model the goal setting process with parents and suggest a general range of age-appropriate dietary and physical activity targets that might be appropriate for each child and parent.

Health Education Condition: Both the child and parent will attend the treatment sessions in this program. This condition will include 23 group meetings on the same schedule as the previously described conditions. Each session will last 90 minutes. The Health Education condition will be tailored for children and families, and will include a series of meetings addressing key aspects of nutrition, physical activity, and health promotion. The health education curriculum will include topics such as national guidelines regarding proper nutrition, guidelines for physical activity, strategies to cope with stress, healthy sources and guidelines for intake of fiber, calcium, protein, grains & carbohydrates. Topics will also include use of vitamin & mineral supplements, dental and sleep hygiene, self-esteem, family communication, and assertiveness training in dealing with peer victimization. The families in the Health Education group will not receive training in behavioral self-regulation strategies, such as goal setting and self-monitoring. Children will participate in a group physical activity during each session such as frisbee, jump rope, stoplight tag. They will also sample healthy snacks such as pretzels or fruits and vegetables. There will be no discussion of implementing these activities and preparing healthy snacks in other settings. Children will not help prepare the snack items.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 8 and 12 years,
* BMI equal to or above the 85th percentile for age and gender
* Child and participating parent(s) or legal guardian(s) are required to live within the same dwelling in a rural county.
* Participating parents or legal guardians must be age 75 years or less.

Exclusion Criteria:

* Child or participating parent has a dietary or exercise restriction
* Medical condition that contraindicates mild energy restriction or moderate physical activity
* Children or adults cannot be engaged in another weight control program.
* Unwilling or unable to give informed consent,
* Parent(s) or legal guardian(s) unable to read English at approximately the 5th grade level,
* Unwilling to accept random assignment,
* Unable to travel to the Extension office for intervention sessions,
* Likely to move out of the county within the next 24 months.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 314 (Actual)
Dates: Start 2009-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Child BMI Z score | 2 years
  Change in Child BMI Z score from baseline to year 2

SECONDARY OUTCOMES:
Child caloric intake | 2 years
  Change in child caloric intake from baseline to year 2.
Child Physical Activity | 2 years
  Change in physical activity from baseline to year 2

CONTACTS AND LOCATIONS:
Overall Officials: David M Janicke, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Janicke DM, Lim CS, Perri MG, Bobroff LB, Mathews AE, Brumback BA, Dumont-Driscoll M, Silverstein JH. The Extension Family Lifestyle Intervention Project (E-FLIP for Kids): design and methods. Contemp Clin Trials. 2011 Jan;32(1):50-8. doi: 10.1016/j.cct.2010.08.002. Epub 2010 Aug 11. PMID 20708715
- [Background] Lim CS, Mayer-Brown SJ, Clifford LM, Janicke DM. Pain is Associated with Physical Activity and Health-Related Quality of Life in Overweight and Obese Children. Child Health Care. 2014 Jul;43(3):186-202. doi: 10.1080/02739615.2013.837825. PMID 25484483
- [Background] Lim, C.S. & Janicke, D.M. (2013). Barriers related to delivering pediatric weight management interventions to children and families from rural communities. Children's Health Care, 42, 214-230.
- [Result] Gowey MA, Lim CS, Clifford LM, Janicke DM. Disordered eating and health-related quality of life in overweight and obese children. J Pediatr Psychol. 2014 Jun;39(5):552-61. doi: 10.1093/jpepsy/jsu012. Epub 2014 Mar 26. PMID 24676798
- [Result] Fedele DA, Janicke DM, Lim CS, Abu-Hasan M. An examination of comorbid asthma and obesity: assessing differences in physical activity, sleep duration, health-related quality of life and parental distress. J Asthma. 2014 Apr;51(3):275-81. doi: 10.3109/02770903.2013.873807. Epub 2014 Jan 10. PMID 24320738
- [Result] Labyak CA, Janicke DM, Lim CS, Colee J, Mathews AE. Anthropometrics to Identify Overweight Children at Most Risk for the Development of Cardiometabolic Disease. Infant Child Adolesc Nutr. 2013 Dec;5(6):341-346. doi: 10.1177/1941406413501379. PMID 25485038
- [Derived] Janicke DM, Lim CS, Perri MG, Mathews AE, Bobroff LB, Gurka MJ, Parish A, Brumback BA, Dumont-Driscoll M, Silverstein JH. Featured Article: Behavior Interventions Addressing Obesity in Rural Settings: The E-FLIP for Kids Trial. J Pediatr Psychol. 2019 Sep 1;44(8):889-901. doi: 10.1093/jpepsy/jsz029. PMID 31039250
- [Derived] Graef DM, Janicke DM, McCrae CS. Sleep patterns of a primarily obese sample of treatment-seeking children. J Clin Sleep Med. 2014 Oct 15;10(10):1111-7. doi: 10.5664/jcsm.4112. PMID 25317092